CLINICAL TRIAL: NCT06080841
Title: Evaluation of Curcumin Supplementation on p53 Levels and Apoptosis in Tumor Cells From Patients With Locally Advanced Cervical Cancer
Brief Title: Curcumin Supplementation in Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Sabinsa Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI/1598/21
Record Dates: First submitted 2023-09-19; First posted 2023-10-12 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: curcumin; locally advanced cervical cancer; p53; apoptosis; chemoradiotherapy
MeSH Terms: interventions — Curcumin; piperine

STUDY DESIGN:
Intervention Model Description: A pilot study in adult women diagnosed with cervical cancer in locally advanced stages (IB3-IVA), who are selected to undergo treatment with concomitant QT-RT followed by BT, by the Functional Gynecology Oncology Unit of the National Cancer Institute.
  The intervention will be supplementation with different doses of curcumin. Patients will eat a standard diet according to their requirements. The aim is to describe the expression of p53 protein levels and apoptosis in tumor cells from these patients. Patients will be monitored by a nutritionist and receive the corresponding care from the medical oncologist.
  Sample size. Because this is a pilot study, the sample size will be at the researcher's convenience; 5 patients per group, 30 patients with locally advanced cervical cancer, who are candidates to receive standard treatment of concomitant chemoradiotherapy, followed by brachytherapy.
  Blood, urine, fecal, and cervicovaginal cytology samples will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (Experimental): 1g of curcumin.
  Interventions: Dietary Supplement: Curcumin
- Group 2 (Experimental): 1 g curcumin + 5 mg piperine.
  Interventions: Dietary Supplement: Curcumin + Piperine
- Group 3 (Experimental): 3 g of curcumin.
  Interventions: Dietary Supplement: Curcumin
- Group 4 (Experimental): 3 g curcumin + 15 mg piperine.
  Interventions: Dietary Supplement: Curcumin + Piperine
- Group 5 (Experimental): 6 g of curcumin.
  Interventions: Dietary Supplement: Curcumin
- Group 6 (Experimental): 6 g curcumin + 15 mg piperine.
  Interventions: Dietary Supplement: Curcumin + Piperine

INTERVENTIONS:
Dietary Supplement: Curcumin — Patients will receive capsules with curcumin C3 (Sabinsa Corp, NJ, USA) containing 1g of curcumin. They will be instructed to consume orally 1 capsule with breakfast for group 1, 1 capsule with each meal for group 3, and 2 capsules with each food for group 5.
  Arms: Group 1; Group 3; Group 5
Dietary Supplement: Curcumin + Piperine — Patients will receive capsules with curcumin C3 (Sabinsa Corp, NJ, USA) containing 1g of curcumin additioned with 5 mg of piperine. They will be instructed to consume orally 1 capsule with breakfast for group 2, 1 capsule with each meal for group 4, and 2 capsules with each meal for group 6.
  Arms: Group 2; Group 4; Group 6

SUMMARY:
Brief Summary.

The goal of this pilot study is to learn about the effect of curcumin supplementation in locally advanced cervical cancer patients. The main questions it aims to answer are:

* Does curcumin supplementation increase the levels of p53 and apoptosis in tumor cells from cervical cancer patients?
* At which dose of curcumin supplementation is the broader effect observed for p53 expression and apoptosis in tumor cells from cervical cancer patients?
* Are all doses safe for supplementation?

Participants will be asked to take curcumin tablets throughout their cancer treatment. Researchers will compare 6 different groups, each group will receive a different dose of curcumin with or without piperin, to see the dose with the broader effect and safety of curcumin supplementation:

1. 1 g of curcumin
2. 1 g of curcumin + piperine
3. 3 g of curcumin
4. 3 g of curcumin + piperine
5. 6 g of curcumin
6. 6 g of curcumin + piperine

DETAILED DESCRIPTION:
BACKGROUND Cervical cancer (CC) continues to be a major public health problem in Mexico. Today more than 4,000 women die each year from this disease, which requires implementing strategies that can improve current treatments, particularly for locally advanced disease. Today it is clear that persistent high-risk Human Papillomavirus infections are the main risk factor for developing CC. At the National Cancer Institute of Mexico (INCan), 80% of patients are diagnosed at locally advanced stages (IB3-IVA). The standard treatment for these stages is concomitant chemoradiotherapy (CCRT) followed by brachytherapy (BT).

p53 restricts tumor growth, promoting cell death and decreasing cell viability. Activation of p53 is vital for CCRT-induced cytotoxicity, while inactivation of p53 has been associated with resistance or insensitivity to treatment. Different nutraceuticals such as berberine and curcumin can reactivate endogenous p53 and exhibit its effects in CC. The E6 oncoprotein inactivates the p53 pathway in CC; therefore, the restoration of p53 may be a promising therapeutic strategy.

The health benefits associated with consuming fruits, vegetables, teas, and spices are due to the presence of phytochemicals. Diets characterized by regular consumption of fruits and vegetables have been associated with a decrease in the risk of CC. A particular group of phytochemicals of interest is polyphenols. The polyphenol curcumin is considered safe and non-toxic by the FDA (Food and Drug Administration), and its administration causes minimal low-grade adverse effects (mainly grade 1 diarrhea). Based on clinical trials' safety and toxicity profile, a dose of up to 8000 mg/day of curcumin can be considered safe.

The current information on the bioavailability of phytochemicals continues to be limited, which places great importance on the exploration of polyphenols as possible new therapeutics. However, the low bioavailability and complex metabolism linked to polyphenols make it difficult to recommend a dose for daily consumption. The addition of piperine to curcumin supplementation has been demonstrated to increase absorption in the intestine.

Different biological effects have been associated with curcumin supplementation in cancer patients. Patients with pancreatic cancer received oral administration of curcumin at a dose of 8 g/day for eight months in combination with gemcitabine, which was well tolerated and showed an improvement in overall survival. Curcumin activity was evaluated in patients with metastatic colon cancer, finding that it was safe and tolerable in combination with FOLFOX.

In locally advanced CC patients, the effect that curcumin has on the expression of p53 in tumor cells has not been investigated, although in vitro studies have demonstrated its effect on the inhibition of oncoproteins, such as E6, and the consequent stabilization of p53, which makes CC cells more susceptible to being destroyed.

The present pilot study seeks to demonstrate that curcumin supplementation will regulate molecular markers, such as p53 and apoptosis in tumor cells, which could provide the basis to study further whether this modulation by curcumin leads to a greater susceptibility of the tumor to standard cancer treatment and, therefore, a better response to treatment.

METHODS The work will be carried out at the National Cancer Institute of Mexico (INCan) in patients with locally advanced CC. Six supplementation groups will be included; in three groups, curcumin will be administered in tablets in oral doses of 1, 3, and 6 g / day respectively, and in the other three groups, curcumin will be administered in tablets in oral doses of 1, 3, and 6 g / day respectively plus 5 mg of piperine/g of curcumin (to facilitate the absorption of curcumin).

Invitation to the study protocol: Diagnosis will be confirmed in the INCan Functional Gynecology Oncology Unit. The corresponding studies are carried out to corroborate that the patient meets the inclusion criteria. On the day of the invitation to the patient, the patient will be explained what the study consists of, and the Informed Consents will be read. If the patient agrees to participate and signs the consent, she will be assigned to the corresponding curcumin dose group.

The patients will be followed for four visits throughout the study: (1) 2 weeks before the beginning of treatment; (2) at the beginning of CRT; (3) at the third cycle of CRT; and (4) at BT.

Patients will be evaluated in 4 visits:

* Visit 1: Indications for a standard diet will be given according to the patient's requirements. Curcumin will be provided to the patient, and instructions for its use will be given according to the group to which she has been assigned. Urine and serum samples will be collected. A cervical swab sample will be obtained.
* Visit 2: The day of initiation of treatment with concomitant CRT. Feces, urine, and serum samples will be collected. A cervical swab sample will be obtained.
* Visit 3: Once the 3 CRT cycles have been completed. Feces, urine, and serum samples will be collected. A cervical swab sample will be obtained.
* Visit 4: When starting treatment with BT. Urine and serum samples will be collected.

Biological samples:

Cervicovaginal cytologies will be taken at each visit. The samples will be analyzed by flow cytometry to quantify p53 positive cells and annexin will be used to identify apoptosis.

Adherence to supplementation will be monitored, bioavailability will be investigated, gastrointestinal toxicity determined, and the safety of supplementation evaluated. Gastrointestinal symptoms will be classified at each visit during treatment according to common toxicity criteria (CTCAE v. 5). Liver function tests, renal function tests, blood chemistry, and hematic biometry will be monitored to assess curcumin supplementation safety. Stool, urine, and serum samples will be taken, from which the bioavailability of curcumin will be assessed by liquid chromatography-electrospray ionization-mass spectrometry. A comparative analysis of these variables will be made between the different supplementation groups to establish the dose in which an impact on the expression of p53 and apoptosis is observed.

Analysis of data:

Data will be analyzed using Statistica software, and graphs will be made in GraphPad Prism. A single-factor repeated measures analysis will be performed with repeated measures across all treatments. The analysis plan will consist of:

* Normality test. The Shapiro-Wilk test will be performed to know if the variables' distribution is normal.
* Descriptive analysis. The distribution of the quantitative independent variables will be determined using the Kolmogorov-Smirnov test. The mean ± standard deviation will be reported for variables with normal distribution or median with 25th and 75th percentiles for variables with free distribution.
* One-way or two-way ANOVA will be performed to determine the significance of differences between groups, followed by Tukey's test for the significance of differences. Confidence intervals will be constructed at 95%, and a value will be declared statistically significant when p is <0.05.
* Multivariate analysis. The following tests will be used to determine if there are differences between the patients who were supplemented with the different doses of curcumin and those who also received piperine:

  * Student's T test for quantitative variables with normal distribution.
  * Mann Whitney U test for quantitative variables with free distribution or ordinal variables.
  * Chi-square test for dichotomous and polytomous variables.

EXPECTED RESULTS AND PERSPECTIVES The investigators expect that curcumin supplementation will stabilize the expression of p53 and increase the apoptosis of tumor cells. The investigators also expect that piperine will increase its absorption. In addition, a dose in humans associated with the expression of p53 has not been reported, so this study will allow the identification of the dose that favors said expression in humans. In addition to its molecular effect, due to its antioxidant properties, the investigators expect that patients will improve gastrointestinal symptoms associated with treatment with CCRT.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding the nature of the study and giving a written consent report.
2. Women > 18 years old.
3. ECOG performance status: 0-2.
4. Be willing and able to comply with scheduled visits, treatment plans, and laboratory tests.
5. Patients with a histological cervical cancer diagnosis: squamous cell, adenosquamous, adenocarcinoma, and glassy cell carcinoma.
6. Classified with clinical stage IB3-IVA (FIGO 2018).
7. Candidates to receive concomitant QT-RT followed by BT.
8. With disease measurable by any imaging method (CT/MRI/PET-CT) according to RECIST v 1.1 criteria.
9. Patients without prior treatment based on QT-RT.
10. Hemoglobin ≥ 10 g/dL.
11. Leukocytes ≥ 4000/mm3.
12. Platelets ≥ 100,000/mm3.
13. Adequate liver function.

Exclusion Criteria:

1. Patients undergoing nutritional treatment or ingesting any dietary supplement, including those containing turmeric or turmeric derivatives, ginger, or rhizome of the turmeric family.
2. Patients with uncontrolled intercurrent diseases, including active infections that contraindicate CT.
3. Patients receiving concomitant treatment with an experimental drug.
4. Patients with vesicovaginal or vesicorectal fistula are diagnosed.
5. Patients with previous or concomitant malignancy except non-melanoma skin carcinoma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
p53 expression | Through study completion, an average of 3 years
  Using the liquid-based cervicovaginal cytology samples, p53 will be quantified by the ELISA method. p53 positive cells will be quantified through flow cytometry.
Frequency of Apoptosis | Through study completion, an average of 3 years
  A conjugate of Annexin V and fluorophore will be used to determine apoptosis in cells from liquid-based cytology, through flow cytometry. The number of apototic cells (positive for Annexin V) will be quantified, and the percentage will be calculated.

SECONDARY OUTCOMES:
Frequency of Gastrointestinal toxicity | Through study completion, an average of 3 years
  Symptoms of gastrointestinal toxicity will be recorded and graded at each visit during treatment according to the common toxicity criteria of adverse events (CTCAE v.5). Frequency and severity will be assessed.
Bioavailability of curcumin | Through study completion, an average of 3 years
  To determine the bioavailability of curcumin, blood, fecal, and urine samples will be obtained. It is proposed to use Chen's method (1997) with some modifications to determine the total amount of bioactive, including lupeol and polyphenols free and in conjugated form; the methodology will depend on the corresponding biological sample, by ultra-high resolution liquid chromatography with chemical ionization at atmospheric pressure coupled or electrospray ionization with MS (UPLC-API or ESI-MS/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Denisse Castro, RDN, PhD, Principal Investigator — Conacyt / National Cancer Institute of Mexico
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The final report will be shared, and other information or data will be shared upon reasonable request.